CLINICAL TRIAL: NCT07330024
Title: Evaluation of Salivary and Pulpal Levels of Substance P and Calcitonin Gene-Related Peptide in Relation to Dental Pain, Pulpal Inflammation, and Psychological Status
Brief Title: Evaluation of Pulpal and Salivary Neuropeptides in Dental Pain
Acronym: PAIN-SPCGRP
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Aliye Kamalak, Assoc. Prof., Kahramanmaras Sutcu Imam University
Other Study IDs: HRÜ/24.15.46; HRÜ/24.15.46 (Other: Harran University Medical Ethics Committee)
Record Dates: First submitted 2025-12-12; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Dental Pain; Pulpitis; Pulpal Inflammation; Psychological Stress; Anxiety
Keywords: Dental Pain; Substance P; Calcitonin Gene-Related Peptide; Saliva Biomarkers; Pulpal Inflammation; Psychological Stress; Anxiety; Depression
MeSH Terms: conditions — Toothache; Pulpitis; Stress, Psychological; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Pulp tissue and unstimulated saliva samples collected during routine endodontic procedures and retained for biochemical analysis of Substance P and Calcitonin Gene-Related Peptide. No DNA extraction is performed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Painful Group: Participants presenting with dental pain who require endodontic treatment and report pain based on clinical examination and Verbal Rating Scale assessment.
- Painless Group: Participants without dental pain who require endodontic treatment and report no pain based on clinical examination and Verbal Rating Scale assessment.

SUMMARY:
This observational cross-sectional study is designed to evaluate pulpal and salivary levels of Substance P (SP) and Calcitonin Gene-Related Peptide (CGRP) in individuals with and without dental pain. The study aims to assess the associations between neuropeptide levels, pain severity, histopathological pulpal inflammation, and psychological status including depression, anxiety, and stress. By integrating biological and psychosocial parameters, this study seeks to contribute to a comprehensive understanding of the multifactorial nature of dental pain.

DETAILED DESCRIPTION:
Dental pain is a multifactorial condition influenced by peripheral inflammatory processes, neurogenic mechanisms, and psychological factors. Neuropeptides such as Substance P (SP) and Calcitonin Gene-Related Peptide (CGRP) are known to play an important role in pain transmission and pulpal inflammatory responses. However, the invasive nature of pulpal sampling limits the routine clinical application of pulpal biomarkers, emphasizing the need to investigate non-invasive biological media such as saliva.

This observational cross-sectional study includes adult participants who require endodontic treatment and are categorized into painful and painless groups based on clinical examination and pain assessment using the Verbal Rating Scale (VRS). Pulp tissue samples are obtained during routine endodontic access procedures, and unstimulated saliva samples are collected before and after the clinical procedure. Levels of SP and CGRP in pulp and saliva samples are measured using enzyme-linked immunosorbent assay (ELISA).

Psychological status is evaluated using the Depression Anxiety Stress Scale-21 (DASS-21) to assess levels of depression, anxiety, and stress. Pulpal inflammation is evaluated through histopathological examination of pulp tissue samples using a semi-quantitative scoring system.

The primary objective of this study is to evaluate the relationship between dental pain and pulpal and salivary neuropeptide levels. Secondary objectives include assessing the associations between neuropeptides, psychological status, pain severity, and histopathological pulpal inflammation. The study is designed to provide descriptive and associative data without intervention, supporting a biopsychosocial framework for understanding dental pain and exploring the potential clinical relevance of salivary biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* ASA physical status I or II
* Presence of permanent teeth requiring endodontic treatment
* Ability to understand the study procedures and provide written informed consent
* No use of analgesic medications within 24 hours prior to clinical assessment
* No food or drink intake within 2 hours prior to saliva sampling

Exclusion Criteria:

* Periodontal disease (probing depth >4 mm or bleeding on probing >20%)
* Systemic inflammatory, autoimmune, neuropathic, or chronic pain disorders
* Acute infection, fever, or antibiotic use within the last 7 days
* Pregnancy or lactation
* Regular use of psychiatric medications (e.g., antidepressants, anxiolytics, antipsychotics, antiepileptics)
* Tobacco use or alcohol consumption within the last 24 hours
* Previous endodontic treatment or history of dental trauma in the study tooth
* Systemic diseases that may affect neuropeptide levels (e.g., diabetes mellitus, thyroid disorders, renal or hepatic disease)
* Use of medications affecting salivary flow

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult individuals aged 18 to 65 years who present to a university dental hospital and require endodontic treatment for permanent teeth. Participants include individuals with dental pain and individuals without dental pain, classified based on clinical examination and pain assessment. All participants are systemically healthy or have ASA physical status I or II and provide written informed consent prior to participation.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Pulpal Calcitonin Gene-Related Peptide (CGRP) Concentration | Periprocedural (single assessment at the time of endodontic access)
  Calcitonin Gene-Related Peptide (CGRP) concentration measured in pulpal tissue samples collected during routine endodontic access. CGRP levels are quantified using enzyme-linked immunosorbent assay (ELISA) and expressed as picograms per milligram of pulp tissue (pg/mg). Higher values indicate increased neurogenic activity and pulpal stress.
Salivary Substance P (SP) Concentration - Baseline | Baseline (prior to clinical procedure)
  Substance P (SP) concentration measured in unstimulated whole saliva samples collected before the clinical procedure. SP levels are analyzed using enzyme-linked immunosorbent assay (ELISA) and expressed as picograms per milliliter (pg/mL). Higher values indicate increased neurogenic and stress-related activity.
Salivary Substance P (SP) Concentration - Periprocedural | Periprocedural (immediately after the clinical procedure; single assessment)
  Substance P (SP) concentration measured in unstimulated whole saliva samples collected immediately after the clinical procedure. SP levels are analyzed using enzyme-linked immunosorbent assay (ELISA) and expressed as picograms per milliliter (pg/mL). Higher values indicate increased neurogenic and stress-related activity.

SECONDARY OUTCOMES:
Dental Pain Severity (Verbal Rating Scale - VRS) | Baseline (at clinical examination prior to treatment)
  Dental pain severity assessed using the Verbal Rating Scale (VRS) with the following categories:
  0 = No pain
  1. = Mild pain
  2. = Moderate pain
  3. = Severe pain
  The scale ranges from 0 to 3, with higher scores indicating greater pain severity.
Psychological Status - Depression Anxiety Stress Scale-21 (DASS-21) | Baseline (at clinical examination prior to treatment)
  Psychological status assessed using the Depression Anxiety Stress Scale-21 (DASS-21), consisting of three subscales: depression, anxiety, and stress.
  Each subscale score ranges from 0 to 42, with higher scores indicating worse psychological status.
Histopathological Pulpal Inflammation Score | Periprocedural (after pulp tissue collection during endodontic access)
  Degree of pulpal inflammation assessed by histopathological examination of pulp tissue samples using a semi-quantitative scoring system:
  0 = No inflammation
  1. = Mild inflammation
  2. = Moderate inflammation
  3. = Severe inflammation
  Higher scores indicate greater inflammatory severity.
Correlation Between Neuropeptide Levels and Psychological Parameters | Baseline (single assessment during study participation)
  Correlation analysis between:
  Pulpal CGRP concentration (pg/mg),
  Salivary Substance P concentration (pg/mL), and
  Psychological parameters (depression, anxiety, stress scores measured by DASS-21).
  Associations are evaluated using appropriate statistical correlation analyses. This outcome does not represent a new biological measurement but an analytical relationship between predefined outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sutcu İmam University, Faculty of Dentistry, Kahramanmaraş, onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) will not be shared due to ethical restrictions, institutional policies, and the sensitive nature of biological and psychological data collected in this study.